CLINICAL TRIAL: NCT01673412
Title: Research of Prognostic Factors Associated With Healing of Venous Leg Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Institut de Recherches Internationales Servier (Other); Société de Dermatologie Française (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AOL02-DR-LOK; 02H37 (Other: CPP Nord-Ouest II)
Record Dates: First submitted 2012-07-31; First posted 2012-08-28 (Estimated); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Leg Ulcer
Keywords: venous leg ulcer healing prognostic factors
MeSH Terms: conditions — Leg Ulcer | interventions — Psychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- interventional arm (Experimental): Psychological tests
  Interventions: Other: Psychological tests

INTERVENTIONS:
Other: Psychological tests — social and economical level intellectual quotient (Raven's Progressive Matrices Standard) Coopersmith self-esteem inventory BECK Depression inventory Minimal Mental Status

SUMMARY:
This study was undertaken to identify prospectively which clinical venous leg ulcer (VLU) characteristics known as possible prognostic markers, and which sociodemographic and psychologic factors associated with VLU are associated with complete healing at 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* ambulatory or hospitalized patients
* patients over 50 years old
* one or more venous leg ulcer, lasting for 1 month or more
* wound area more than 1 cm2
* clinical findings consistent with established venous disease (skin hyperpigmentation, varicose veins, lipodermatosclerosis), confirmed by venous Doppler duplex ultrasonography performed during the preceding 6 months
* absence of significant arterial insufficiency assessed by clinical findings (intermittent claudication or resting pain, necrotic or distal foot wound) and by an ankle brachial index (ABI) ≥0.8
* ability to give informed consent
* ability to be followed for 24 weeks

Exclusion Criteria:

* ongoing systemic diseases known to be associated with pyoderma gangrenosum or necrotizing vasculitis
* corticosteroid, cytotoxic or immunosuppressant drug use during the preceding 3 months
* hypertensive leg ulcer
* foot ulcer
* ABI < 0.8

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2003-01; Primary Completion 2008-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Healing or non-healing of venous leg ulcers at week 24 | week 24
  Healing or non-healing of venous leg ulcers at week 24

SECONDARY OUTCOMES:
clinical characteristics | week 24
  comparison between healed and non healed venous leg ulcers at week 24 for patient clinical characteristics (age, weight, body mass index, concomitant diseases, medical and surgical history, autonomy, mobility)
biologic characteristics | week 24
  comparison between healed and non healed venous leg ulcers at week 24 for patient biologic characteristics (complete blood count, hemoglobinemia, albuminemia, and only for patients with diabetes mellitus : glycemia and glycated haemoglobin)
psychologic assessments | week 24
  comparison between healed and non healed venous leg ulcers at week 24 for patient psychologic assessments (self-esteem assessed by Coopersmith self-esteem inventory, symptoms of depression researched with Beck Depression Inventory)
cognitive assessments | week 24
  comparison between healed and non healed venous leg ulcers at week 24 for patient cognitive assessments (intellectual quotient evaluated by Raven's progressives matrices test, signs of intellectual deterioration assessed by Minimal Mental Status test)
social assessment | week 24
  comparison between healed and non healed venous leg ulcers at week 24 for patient social assessments (assessment of social and occupational group, of education level, of income level and of marital status)
affected-leg characteristics | week 24
  comparison between healed and non healed venous leg ulcers at week 24 for patient affected-leg inclusion characteristics (venous insufficiency classified using CEAP classification, ultrasonography assessment of leg with measurement of the Ankle Brachial Index (ABI) and examination of the leg venous system, number of ulcers on target leg, presence/absence of venous abnormalities (varicose veins, ochre dermatitis, white atrophy, acute hypodermitis), of cutaneous signs of lymphatic insufficiency, of oedema and of ankle articulation ankylosis)
venous leg ulcers inclusion characteristics | week 24
  comparison between healed and non healed venous leg ulcers at week 24 for patient venous leg ulcers inclusion characteristics (size, localization, duration, percentage of granulation/fibrinous tissue, aspect of ulcer's margins, pain)
venous insufficiency treatment | week 24
  comparison between healed and non healed venous leg ulcers at week 24 for patient venous insufficiency treatment (compliance to venous contention assessed by an evaluating questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine LOK, PhD, Principal Investigator — Centre Hospitalo-Universitaire d'Amiens
Locations (35):
- France (35):
  - Centre Hospitalo-Universitaire d'Amiens - Dermatologie, Amiens
  - Hôpital Saint Vincent de Paul - Médecine interne et Gériatrie I, Amiens
  - Hôpital Victor Dupouy - Dermatologie, Argenteuil
  - Hôpital Saint Jacques - Dermatologie 1, Besançon
  - CHU de Brest - Dermatologie, Brest
  - CHU Clémenceau - Dermatologie, Caen
  - Hôpitaux Civils de Colmar - Service de Dermatologie, Colmar
  - CHU Bocage - Dermatologie, Dijon
  - CHU Michallon - Dermatologie, Grenoble
  - Hôpital C. Foix - Service de Gérontologie, Ivry
  - Centre Hospitalier - Service de Médecine Interne, Lens
  - Hôpital Robert Boulin - Dermatologie, Libourne
  - Hôpital Claude Huriez - Clinique Dermatologique, Lille
  - CHRU Dupuytren - Dermatologie, Limoges
  - Hôpital Saint Philibert - Dermatologie, Lomme
  - Hôpital d'Instruction des Armées Desgenettes, Lyon
  - Hôpital Sainte Marguerite - Dermatologie, Marseille
  - Hôpital SAint Charles - Dermatologie, Montpellier
  - Hôpital Fournier, Nancy
  - Hôpital Rothschild - Consultation de Dermatologie, Paris
  - CHU Bichat - Service de Dermatologie, Paris
  - Hôpital Saint Louis - Service de Dermatologie, Paris
  - Hôpital Broussais - Rééducation Vasculaire, Paris
  - Hôpital du Haut Levêque - Dermatologie, Pessac
  - Centre Hospitalier Laennec - Dermatologie, Quimper
  - CHU Robert Debré, Reims
  - CHU Pontchaillou, Rennes
  - Cabinet de Dermatologie 43, rue Jean Lecanuet, Rouen
  - Hôpital Charles NICOLLE - Service de Dermatologie, Rouen
  - Le Royal Parc - Dermatologie, Saint-Brieuc
  - Centre Hospitalier Intercommunal Poissy Saint Germain, Saint-Germain-en-Laye
  - Cabinet de Dermatologie 1,rue dembarrère, Tarbes
  - Hôpital Beauregard, Thionville
  - CHU Trousseau - Dermatologie, Tours
  - Centre Hospitalier de Valence - Dermatologie, Valence

REFERENCES:
- [Result] Chaby G, Senet P, Ganry O, Caudron A, Thuillier D, Debure C, Meaume S, Truchetet F, Combemale P, Skowron F, Joly P, Lok C; Angio-Dermatology Group of the French Society of Dermatology. Prognostic factors associated with healing of venous leg ulcers: a multicentre, prospective, cohort study. Br J Dermatol. 2013 Nov;169(5):1106-13. doi: 10.1111/bjd.12570. PMID 23909381